CLINICAL TRIAL: NCT05027568
Title: Randomized, Double-blind, Placebo-controlled, Dose Escalation Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of IOA-289 in Healthy Male Volunteers
Brief Title: A Study to Assess an ATX Inhibitor (IOA-289) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOA-289-101
Record Dates: First submitted 2021-07-16; First posted 2021-08-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Healthy subjects, effect of food, Roginolisib
MeSH Terms: interventions — Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IOA-289 daily oral dosing plus gemcitabine and nabpaclitaxel every 3 weeks starting on Day 8 (Experimental)
  Interventions: Drug: IOA-289; Drug: Nab paclitaxel / gemcitabine

INTERVENTIONS:
Drug: IOA-289 — Daily oral twice daily dosing of IOA-289
Drug: Nab paclitaxel / gemcitabine — Given in combination with IOA-289

SUMMARY:
The purpose of Part 1 of this First-in-Human trial is to evaluate the safety and tolerability after single ascending oral doses of IOA-289 given to healthy male subjects, compared to placebo. After the oral dose administrations, the amount of IOA-289 present in serum will be determined for pharmacokinetic characterisation. Also the reduction of LPA in plasma will be determined as a pharmacodynamic biomarker.

Part 2 is optional and its conduct will be dependent on the pharmacokinetic data generated in Part 1. Part 2 will be a randomized, crossover, open label, single oral dose administration of IOA-289 to healthy male subjects either in a fasted state, or after a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 50 years of age (inclusive) at the screening visit
* Body mass index between 18.0 and 30.0 kg/m2 (inclusive) at the screening visit
* In good health as determined by medical history, physical examination, ECG, serum/urine, clinical chemistry, haematology, and serology tests
* Able to provide written, informed consent prior to initiation of any trial-related procedures, and able, in the opinion of the Principal Investigator, to comply with all the requirements of the trial
* Male subjects who are surgically sterile (i.e., have undergone bilateral orchidectomy); and male subjects who agree to remain abstinent or to practice double-barrier forms of birth control and refrain from sperm donation from trial screening through 90 days from the last dose of IMP

Exclusion Criteria:

* Clinically significant abnormality in past medical history, or at the screening physical examination, that in the Investigator's or Sponsor's opinion may place the subject at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of IMP
* History of drug and/or alcohol abuse within 2 years prior to the screening visit
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of HBsAg, anti-HCV, and/or HIV antibodies
* History of any significant drug allergy
* Positive alcohol breath test and/or urine drug screen for substance of abuse at the screening visit or upon check-in to the clinical trial site
* History of having taken an investigational drug within 30 days preceding trial entry
* History of significant bleeding or haemorrhagic tendencies
* Donation of blood or plasma within 30 days prior to dosing
* Use of prescription medication, over-the-counter medication, herbal medication, or vitamin supplements within 14 days prior to dosing and antibiotics within 30 days prior to dosing. The Sponsor may allow exceptions only if the medication's administration is deemed unlikely to impact the PK result
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to screening (e.g., occupational exposure to pesticides, organic solvents)
* Supine blood pressure, after resting for ≥3 minutes, higher than 140/90 mmHg or lower than 100/50 mmHg. The Sponsor may allow exceptions if they are not deemed clinically significant
* Supine pulse rate, after resting for ≥3 minutes, outside the range of 50 to 90 bpm. The Sponsor may allow exceptions if they are not deemed clinically significant
* History of serious mental disorders that, in the opinion of the Investigator, would exclude the subject from participating in this trial

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Numbers of participants with treatment-related adverse events as assessed by MedDRA v24 | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  Adverse Events will be assessed by nondirective questioning of the participants during the screening process and at each visit during the study

SECONDARY OUTCOMES:
Pharmacokinetic profile of IOA-289 | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  Blood samples for plasma IOA-289 concentrations
Cmax | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  The maximum observed plasma concentration
Tmax | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  The time at which Cmax occurs
AUCinf | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  The area under the plasma concentration-time curve from time of dosing to infinity
To determine the change from baseline of LPA levels | Day 1: Predose and at 0.5,1, 2, 4, 8, 10 and 24 hours postdose
  Measurement of LPA levels in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Ricerche Cliniche di Verona srl, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No